CLINICAL TRIAL: NCT01853410
Title: Peripheral Stimulation Device to Improve Coronary Flow Reserve in Coronary Artery Disease
Acronym: PERCCAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 103661
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Ischemic Disease
Keywords: coronary artery disease; coronary flow reserve; endothelial function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gekoTM device application (Experimental): Single arm study. Application of gekoTM device as described above with assessment of effect on coronary flow and endothelial function.
  Interventions: Device: gekoTM

INTERVENTIONS:
Device: gekoTM

SUMMARY:
The purpose of the PERCCAD Study is to investigate the effect of the gekoTM device (a non-invasive calf muscle stimulator approved for use to improve blood flow by Health Canada) on coronary blood flow in order to assess its potential role as a therapeutic modality for the treatment of symptomatic coronary artery disease (CAD). This will occur in patients already undergoing coronary angiography and percutaneous coronary intervention (PCI) as part of their usual medical care. Further, the investigators will also assess the overall effect on blood flow in the body using non-invasive techniques. The primary objective of the PERCCAD study is to assess the effect of the gekoTM device on coronary blood flow in patients with symptomatic CAD who are undergoing invasive angiographic assessment and management with PCI. This evaluation of the gekoTM device is to be performed at the time of the patient's already planned invasive assessment and management so that invasive data can be collected without exposing the patient to risks other than those already associated with their planned procedure and usual clinical care. The secondary objective of the study is to assess the effect of muscle stimulation with the gekoTM device on endothelial function and peripheral blood flow measured via non-invasive techniques.

DETAILED DESCRIPTION:
Angina pectoris or anginal equivalent dyspnoea are frequent symptoms related to impaired myocardial blood supply. The supply-demand imbalance that arises in the setting of coronary artery disease can be addressed by improving myocardial blood supply through mechanical revascularization with percutaneous coronary intervention or bypass surgery or by reducing myocardial energy demand through pharmacotherapy including the use of negative chronotropic agents such as beta blockers. When further revascularization is not an option, or standard therapies are insufficient to control symptoms, other novel therapies are attempted to improve myocardial blood supply and decrease angina. Enhanced external counterpulsation (EECP) devices have been demonstrated to augment cardiac performance and coronary flow and have a beneficial effect in reducing anginal symptoms in patients with CAD.(1-4) Transcutaneous (non-invasive) electrical nervous stimulation of skeletal muscle to improve venous return to the heart and provide a potential mechanism to augment and improve blood flow, including coronary flow, is a potential alternative method to achieve a similar effect,(5,6) but is less cumbersome and more easily integrated into clinical practice. The gekoTM device is a small transcutaneous nerve stimulator (weight 18g, dimensions 149mm x 42mm x 11mm) that is applied non-invasively to the skin over the common peroneal nerve in the lower limb that has been demonstrated to safely stimulate blood flow from the gastrocnemius and soleus venous system via activation of the venous 'pump' system, intrinsic to the calf muscles. As a result, the gekoTM device is approved for use in Canada to improve blood flow and is already being used in clinical practice at University Hospital. By improving venous return, this device has the potential to have a therapeutic effect in the management of CAD by augmenting coronary blood flow. The purpose of the PERCCAD Study is to investigate the effect of the gekoTM device on coronary blood flow in order to assess its potential role as a therapeutic modality for the treatment of symptomatic CAD. Further, since previous studies with EECP also demonstrated improvement in endothelial function, the investigators plan to study the effect of the gekoTM device on endothelial function and peripheral blood flow in the same patients via non invasive techniques(4, 7, 8) given the established relationship between endothelial dysfunction and cardiovascular risk. (9-12)

The primary objective of the PERCCAD study is to assess the effect of the gekoTM device on coronary blood flow in patients with symptomatic CAD who are undergoing invasive angiographic assessment and management with PCI. This evaluation of the gekoTM device is to be performed at the time of the patient's already planned invasive assessment and management so that invasive data can be collected without exposing the patient to risks other than those already associated with their planned procedure and usual clinical care. The secondary objective of the study is to assess the effect of muscle stimulation with the gekoTM device on endothelial function and peripheral blood flow measured via non-invasive techniques.

Study Design:

Single arm clinical study where patients act as their own controls (coronary flow reserve and endothelial function measured in patients already undergoing angiography and PCI) with measurements recorded pre and post application of the gekoTM device.

Coronary flow assessment: The PCI procedure will be performed according to standard practice. As part of routine practice, a guidewire is inserted into the coronary artery and used as a "rail" for delivering balloons and stents. Often, we use a special Doppler guidewire with a sensor at the tip that is used for measurements of blood flow. We will use such a guidewire for the current study (13-16). Velocity signals are obtained by the guidewire and average peak velocity (APV) is determined. Intracoronary adenosine will be given to induce hyperemia and increase coronary flow (17-21). Intracoronary adenosine is used routinely during PCI. Coronary flow reserve (CFR) will be calculated as the ratio of APV during hyperemia compared to APV at baseline. After measurement of baseline APV and CFR, we will perform two minutes of muscle stimulation using the gekoTM device at a low pulse width setting and record APV. After this, a further two minutes of muscle stimulation using the gekoTM device at a higher pulse width setting will occur with repeated APV and CFR measurements recorded. This process will be performed in at least two coronary arteries at the time of patient's usual invasive assessment and management. Calf muscle stimulation with the gekoTM device: The gekoTM device will be fitted bilaterally behind the patient's knees in the popliteal fossa. At the appropriate time the device will be set to stimulate the common peroneal nerve transcutaneously (the low setting will be set at the level at which the patient has a sensation of stimulation but where there is no visible movement of the lower leg; the high setting will be at the patient's highest tolerable level, but not lower than the level which elicited slight visible movement of the lower leg).

Endothelial Function Assessment: Endothelial function study will be performed on a separate visit following the PCI, by measurement of peripheral vasodilator response using fingertip pulse amplitude tonometry (peripheral arterial tonometry-PAT). PAT signals will be obtained with the EndoPAT2000 (EndoPAT) device (Itamar Medical Inc., Caesarea, Israel). The EndoPAT is an FDA approved device for noninvasive assessment of endothelial dysfunction, it is widely used for clinical and research purposes and validated as a method of endothelial function assessment.(22-24) Specially designed finger probes are placed on the index finger of each patient's hand. The probes are comprised of a system of inflatable latex air cuffs connected by pneumatic tubes to an inflating device controlled through a computer algorithm. There is no occlusion of arterial blood flow. Pulsatile volume changes of the distal digit induce pressure alterations in the finger cuff, which are sensed by pressure transducers and transmitted to and recorded by the EndoPAT. Endothelial function is measured via a reactive hyperemia-peripheral arterial tonometry index (RH-PAT index). A reactive hyperemia protocol consists of a 5-minute baseline measurement, after which a blood pressure cuff placed on the test arm is inflated to 60 mmHg above baseline systolic blood pressure, or at least 200 mmHg for 5 minutes. After 5 minutes, the cuff is deflated, and the PAT tracing recorded for a further 5 minutes. The ratio of the PAT signal after cuff release, compared to baseline, is calculated through a computer algorithm automatically normalizing for baseline signal, and indexed to the contra lateral arm. The calculated ratio reflects the RH-PAT index, a reflection of degree of endothelial function. This process is non-invasive and does not require percutaneous vascular access. Endothelial function will also be assessed at baseline and following 1 hour treatment with the gekoTM using the EndoPAT to calculate the RH-PAT index as described. In addition, the effect on popliteal artery vessel diameter and Doppler flow velocity will also be recorded using a surface ultrasound probe at baseline and following 1 hour of treatment with the gekoTM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80.
2. Symptomatic coronary artery disease and already undergoing invasive angiographic assessment and percutaneous coronary intervention.

Exclusion criteria:

1. Significant valvular heart disease or left ventricular dysfunction.
2. Contraindication to the administration of intracoronary adenosine.
3. Latex allergy.
4. Significant peripheral motor neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Coronary Flow Reserve following stimulation with gekoTM device | Time = 0; Time = post 120 sec stimulation (low setting); Time = post 120 sec stimulation (high setting)
  The change in the effect of the gekoTM device on coronary blood flow as measured by coronary flow reserve using a Doppler tipped coronary flow wire inserted into the coronary artery tree via a percutaneous technique, will be measured at baseline, after 120 sec of stimulation with the gekoTM device on low frequency setting, and after 120 sec of stimulation with the gekoTM device on high frequency setting

SECONDARY OUTCOMES:
Change in Popliteal artery vessel diameter following 60 mins stimulation with gekoTM device | Time = 0; Time = post 60 mins stimulation with gekoTM device
  Change in popliteal artery vessel diameter will be recorded using a surface ultrasound probe at baseline and following 60 mins of treatment with the gekoTM.
  This study will be performed on a separate visit following the PCI procedure.
Change in Popliteal artery vessel Doppler flow velocity following 60 mins stimulation with gekoTM device | Time = 0; Time = post 60 mins stimulation with gekoTM device
  Change in popliteal artery vessel Doppler flow velocity will be recorded using a surface ultrasound probe at baseline and following 60 mins of treatment with the gekoTM. This study will be performed on a separate visit following the PCI procedure.
Change in Endothelial function following 60 mins stimulation with gekoTM device | Time = 0; Time = post 60 mins stimulation with gekoTM device
  The change in Endothelial function study will by measured using the EndoPAT2000 following 60 mins of treatment with the gekoTM. This study will be performed on a separate visit following the PCI procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Loh PH, Cleland JG, Louis AA, Kennard ED, Cook JF, Caplin JL, Barsness GW, Lawson WE, Soran OZ, Michaels AD. Enhanced external counterpulsation in the treatment of chronic refractory angina: a long-term follow-up outcome from the International Enhanced External Counterpulsation Patient Registry. Clin Cardiol. 2008 Apr;31(4):159-64. doi: 10.1002/clc.20117. PMID 18404725
- [Background] Masuda D, Nohara R, Hirai T, Kataoka K, Chen LG, Hosokawa R, Inubushi M, Tadamura E, Fujita M, Sasayama S. Enhanced external counterpulsation improved myocardial perfusion and coronary flow reserve in patients with chronic stable angina; evaluation by(13)N-ammonia positron emission tomography. Eur Heart J. 2001 Aug;22(16):1451-8. doi: 10.1053/euhj.2000.2545. PMID 11482918
- [Background] Michaels AD, Accad M, Ports TA, Grossman W. Left ventricular systolic unloading and augmentation of intracoronary pressure and Doppler flow during enhanced external counterpulsation. Circulation. 2002 Sep 3;106(10):1237-42. doi: 10.1161/01.cir.0000028336.95629.b0. PMID 12208799
- [Background] Yang DY, Wu GF. Vasculoprotective properties of enhanced external counterpulsation for coronary artery disease: beyond the hemodynamics. Int J Cardiol. 2013 Jun 5;166(1):38-43. doi: 10.1016/j.ijcard.2012.04.003. Epub 2012 May 4. PMID 22560950
- [Background] Jawad H. The effect of a novel electrical stimulation method for improving lower limb blood flow in healthy volunteers. 2012
- [Background] Tucker A, Maass A, Bain D, Chen LH, Azzam M, Dawson H, Johnston A. Augmentation of venous, arterial and microvascular blood supply in the leg by isometric neuromuscular stimulation via the peroneal nerve. Int J Angiol. 2010 Spring;19(1):e31-7. doi: 10.1055/s-0031-1278361. PMID 22477572
- [Background] Akhtar M, Wu GF, Du ZM, Zheng ZS, Michaels AD. Effect of external counterpulsation on plasma nitric oxide and endothelin-1 levels. Am J Cardiol. 2006 Jul 1;98(1):28-30. doi: 10.1016/j.amjcard.2006.01.053. Epub 2006 May 3. PMID 16784915
- [Background] Bonetti PO, Barsness GW, Keelan PC, Schnell TI, Pumper GM, Kuvin JT, Schnall RP, Holmes DR, Higano ST, Lerman A. Enhanced external counterpulsation improves endothelial function in patients with symptomatic coronary artery disease. J Am Coll Cardiol. 2003 May 21;41(10):1761-8. doi: 10.1016/s0735-1097(03)00329-2. PMID 12767662
- [Background] Rubinshtein R, Kuvin JT, Soffler M, Lennon RJ, Lavi S, Nelson RE, Pumper GM, Lerman LO, Lerman A. Assessment of endothelial function by non-invasive peripheral arterial tonometry predicts late cardiovascular adverse events. Eur Heart J. 2010 May;31(9):1142-8. doi: 10.1093/eurheartj/ehq010. Epub 2010 Feb 24. PMID 20181680
- [Background] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Menzoian JO, Vita JA. Risk stratification for postoperative cardiovascular events via noninvasive assessment of endothelial function: a prospective study. Circulation. 2002 Apr 2;105(13):1567-72. doi: 10.1161/01.cir.0000012543.55874.47. PMID 11927524
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169
- [Background] Gould KL, Lipscomb K. Effects of coronary stenoses on coronary flow reserve and resistance. Am J Cardiol. 1974 Jul;34(1):48-55. doi: 10.1016/0002-9149(74)90092-7. No abstract available. PMID 4835753
- [Background] Hoffman JI. Maximal coronary flow and the concept of coronary vascular reserve. Circulation. 1984 Aug;70(2):153-9. doi: 10.1161/01.cir.70.2.153. No abstract available. PMID 6234109
- [Background] Collins P. Coronary flow reserve. Br Heart J. 1993 Apr;69(4):279-81. doi: 10.1136/hrt.69.4.279. No abstract available. PMID 8489855
- [Background] Wilson RF, Johnson MR, Marcus ML, Aylward PE, Skorton DJ, Collins S, White CW. The effect of coronary angioplasty on coronary flow reserve. Circulation. 1988 Apr;77(4):873-85. doi: 10.1161/01.cir.77.4.873. PMID 2964950
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Casella G, Leibig M, Schiele TM, Schrepf R, Seelig V, Stempfle HU, Erdin P, Rieber J, Konig A, Siebert U, Klauss V. Are high doses of intracoronary adenosine an alternative to standard intravenous adenosine for the assessment of fractional flow reserve? Am Heart J. 2004 Oct;148(4):590-5. doi: 10.1016/j.ahj.2004.04.008. PMID 15459587
- [Background] Murtagh B, Higano S, Lennon R, Mathew V, Holmes DR Jr, Lerman A. Role of incremental doses of intracoronary adenosine for fractional flow reserve assessment. Am Heart J. 2003 Jul;146(1):99-105. doi: 10.1016/S0002-8703(03)00120-0. PMID 12851614
- [Background] Jeremias A, Whitbourn RJ, Filardo SD, Fitzgerald PJ, Cohen DJ, Tuzcu EM, Anderson WD, Abizaid AA, Mintz GS, Yeung AC, Kern MJ, Yock PG. Adequacy of intracoronary versus intravenous adenosine-induced maximal coronary hyperemia for fractional flow reserve measurements. Am Heart J. 2000 Oct;140(4):651-7. doi: 10.1067/mhj.2000.109920. PMID 11011341
- [Background] Zijlstra F, Juilliere Y, Serruys PW, Roelandt JR. Value and limitations of intracoronary adenosine for the assessment of coronary flow reserve. Cathet Cardiovasc Diagn. 1988;15(2):76-80. doi: 10.1002/ccd.1810150203. PMID 3180211
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Kuvin JT, Mammen A, Mooney P, Alsheikh-Ali AA, Karas RH. Assessment of peripheral vascular endothelial function in the ambulatory setting. Vasc Med. 2007 Feb;12(1):13-6. doi: 10.1177/1358863X06076227. PMID 17451088
- [Background] Hamburg NM, Benjamin EJ. Assessment of endothelial function using digital pulse amplitude tonometry. Trends Cardiovasc Med. 2009 Jan;19(1):6-11. doi: 10.1016/j.tcm.2009.03.001. PMID 19467447